CLINICAL TRIAL: NCT01465360
Title: Performance of AclarusDx™, A Blood-Based Transcriptomic Test for Alzheimer's Disease, in US-based Patients Suffering From Memory Impairment and Newly Referred to A Reference Memory Center, for AD Diagnostic Workup-A Pilot Descriptive Study
Brief Title: Performance of AclarusDx™, a Blood-Based Transcriptomic Test for AD, in US Patients Newly Referred to a Memory Center
Status: Completed | Type: Observational
Sponsor: Exonhit (Industry)
Responsible Party: Sponsor
Other Study IDs: EHTAD/003
Record Dates: First submitted 2011-10-28; First posted 2011-11-04 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Vascular Dementia; Fronto-temporal Dementia; Primary Progressive Aphasia; Parkinson' Disease Dementia; Mixed Dementia
Keywords: Alzheimer's disease; AD; Non AD dementia; Mild Cognitive Impairment; MCI; Vascular dementia; Fronto-temporal dementia; Primary progressive aphasia; Parkinson's Disease dementia; Mixed dementia; Blood signature; Diagnosis; AclarusDx; Alzheimer's Disease and other non-AD dementia; Exonhit
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia, Vascular; Aphasia, Primary Progressive; Mixed Dementias; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood samples collected in PAXgene® blood RNA tubes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study patients: Patients newly referred to a Reference Memory Center with a complaint of memory impairment for AD diagnostic workup.

SUMMARY:
The purpose of this study is to assess the performance of AclarusDx™, an investigational blood test detecting gene expression information, and intended to help physicians in making an Alzheimer's Disease diagnosis in patients having memory impairments.

DETAILED DESCRIPTION:
The objective of this study is to apply AclarusDx™ signature in a reference US Center in 160 patients newly referred to one of the three study centers within the Cleveland Clinic, Center for Brain Health network, for diagnostic workup. Only AclarusDx™ will be added to the panel of tests usually performed at the centers to establish diagnosis. AclarusDx™ will be used for investigational use only, not for diagnostic purpose. The ultimate goal is to define the clinical utility of AclarusDx™ to provide Primary Care Physicians (PCPs) with a tool that will help them in making the diagnosis of Alzheimer's Disease (AD).

The primary objectives are :

1. To obtain an estimate of the capability of AclarusDx™ to identify AD patients among a US-based population of newly referred patients suffering from objective memory impairment which maybe potentially related to multiple and different etiologies.
2. To compare the performance of AclarusDx™ in a US-based population of newly referred patients with memory impairment with the performance of AclarusDx™ observed in one comparable European population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient referred to the center for memory impairment.
* The memory impairment has previously been observed by a caregiver or documented by a physician.
* The memory impairment is confirmed by the memory center.
* Caucasian ethnicity.
* A written informed consent approved by an ethical review board or similar body must be obtained from the patient prior to any study-related procedures.
* If applicable, standard treatment with cholinesterase inhibitor and/or memantine is acceptable.
* Patient estimated to be compliant with study procedures.
* Patient has a level of understanding sufficient to agree to all procedures required by the protocol and must be able to cooperate. Under no circumstances will a subject who does not understand the procedure, be allowed to consent to the procedure.

Exclusion Criteria:

* Recent acute pathology or medical condition or surgery which may alter the inflammatory homeostasis, according to the opinion of the investigator.
* Non-Caucasian ethnicity.
* Patient with severe uncontrolled or unstable medical condition.
* Need for a legal representative for the medical condition of the patient.
* Any current pathology or medical condition, for which blood sampling may involve a risk for the patient's health, according to the opinion of the investigator.
* Current or recent history (within one month) of clinically significant pathology, medical condition (including hospitalization) or symptoms. However, chronic diseases or medical conditions that are considered stable are accepted, provided that they are compatible with other study selection criteria.
* Current or recent history of drug or alcohol abuse or dependence.
* Current, clinically significant major psychiatric disorder (eg, major depressive disorder) according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition text revised (DSM-IV TR), or significant symptoms (eg, hallucinations).
* Woman of childbearing potential is not allowed to participate in the study. (A woman of childbearing potential is a woman who is biologically capable of becoming pregnant).
* Current participation in another study using an investigational non-marketed product.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian patients that are newly referred to a Reference Memory Center with a complaint of memory impairment will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-11

PRIMARY OUTCOMES:
Sensitivity of AclarusDx™ in AD patients | Outcome measured during one single study visit
  The determination of the sensitivity of the test, being the percentage of positive AclarusDx™ calls among referred patients being confirmed clinically as having AD at the Memory Center will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Charles B. Bernick, MD, Principal Investigator — Cleveland Clinic Lou Ruvo Center for Brain Health
Locations (3):
- United States (3):
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Cleveland Clinic Center for Brain Health - Mellen Center, Cleveland, Ohio
  - Cleveland Clinic Senior Care Assessment - Lakewood Hospital, Lakewood, Ohio